CLINICAL TRIAL: NCT05282758
Title: Part 1. Effects of Free Movement Dance as a Physiotherapy Intervention for Female Patients Diagnosed With Chronic Widespread Pain Including (Fibromyalgia) - Prospective Randomised Controlled Trial. Part 2. Exploring the Processes of Free Movement Dance as a Physiotherapy Intervention for Female Patients Diagnosed With Chronic Widespread Pain (Including Fibromyalgia) Over Time - a Qualitative Study. Part 3. Exploring Withdrawal From Study Participation - a Qualitative Study
Brief Title: Effects of and Exploring the Processes of Free Movement Dance as a Physical Therapy Intervention for Female Patients Diagnosed With Chronic Widespread Pain (Including Fibromyalgia).
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPM Dnr: 2021-04146
Record Dates: First submitted 2021-12-20; First posted 2022-03-16 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Fibromyalgia; Chronic Widespread Pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interdisciplinary team treatment + add on Intervention - Free Movement Dance (Experimental): Interdisciplinary team treatment + add on Intervention - Free Movement Dance as a physiotherapy intervention
  Interventions: Other: Free Movement Dance
- Interdisciplinary team treatment + add on Modified person-centered progressive resistance exercise (Active Comparator): Interdisciplinary team treatment + add on Control group - modified person-centered progressive resistance exercise as a physiotherapy intervention
  Interventions: Other: Modified person-centred progressive resistance exercise

INTERVENTIONS:
Other: Free Movement Dance — Free Movement Dance as a physiotherapy intervention
  Arms: Interdisciplinary team treatment + add on Intervention - Free Movement Dance
Other: Modified person-centred progressive resistance exercise — Modified person-centered progressive resistance exercise as a physiotherapy intervention
  Arms: Interdisciplinary team treatment + add on Modified person-centered progressive resistance exercise

SUMMARY:
The study has three parts:

Part 1: To evaluate, for adult female patients diagnosed with chronic widespread pain (including fibromyalgia), the effects of Free Movement Dance as an add-on intervention after interdisciplinary pain management/rehabilitation at a specialist pain clinic versus modified person-centered progressive resistance exercise. The cognitive-behavioural conceptualization of pain, effects on pain intensity, physical function, self-efficacy, pain catastrophizing, health related quality of life, anxiety and depression symptoms and quality of sleep will be evaluated.

Part 2: To explore, for adult female patients diagnosed with chronic widespread pain (including fibromyalgia), the processes of Free Movement Dance, as an add-on intervention after interdisciplinary pain management/rehabilitation at a specialist pain clinic, to generate a substantive theory useful for clinical praxis.

Part 3: To explore and describe why participants who agreed and signed consent choose to withdraw from participating in the interventions of the study's part 1.

ELIGIBILITY:
Inclusion Criteria:

* Female Patients Diagnosed With Chronic Widespread Pain (Including Fibromyalgia) participating in an interdisciplinary pain management and rehabilitation for three months on a specialist pain clinic in south-west of Sweden.
* Age over 18 years and to be able to read and write Swedish. -

Exclusion Criteria:

* Red flag disorders such as malignancy/cancer, acute traumas such as fracture (less than six months ago) or infection.
* Pregnancy, severe mental illness, and ongoing substance abuse.
* Yellow flags as issues with compensation system or unsolved insurance issues with insurance company or the Swedish Social Insurance Agency. -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Cognitive-behavioural conceptualization of pain | Before and after the three months of interdisciplinary specialist interventions and after 12 months, which is standard procedure + after ending the add-on interventions and 24 months after the interdisciplinary treatments
  - measured with The Multidimensional Pain Inventory- Swedish (MPI-s)

SECONDARY OUTCOMES:
Self-reported Pain | Before and after the three months of interdisciplinary specialist interventions and after 12 months, which is standard procedure + after ending the add-on interventions and 24 months after the interdisciplinary treatments
  measured by Numeric Pain Rating Scale (NPRS)
Health Related Quality of Life | Before and after the three months of interdisciplinary specialist interventions and after 12 months, which is standard procedure + after ending the add-on interventions and 24 months after the interdisciplinary treatments
  - Physical function, Physical role and Quality of life measured by Rand - 36
Self-efficacy | Before and after the three months of interdisciplinary specialist interventions and after 12 months, which is standard procedure + after ending the add-on interventions and 24 months after the interdisciplinary treatments
  measured by The General Self-Efficacy Scale (GSE)
Pain catastrophizing | Before and after the three months of interdisciplinary specialist interventions and after 12 months, which is standard procedure + after ending the add-on interventions and 24 months after the interdisciplinary treatments
  measured by the Pain Catastrophizing Scale (PCS)
Health Related Quality of Life | Before and after the three months of interdisciplinary specialist interventions and after 12 months, which is standard procedure + after ending the add-on interventions and 24 months after the interdisciplinary treatments
  measured by the EuroQol-5 dimensions (EQ-5D-3L)
Anxiety and depression symptoms | Before and after the three months of interdisciplinary specialist interventions and after 12 months, which is standard procedure + after ending the add-on interventions and 24 months after the interdisciplinary treatments
  measured by the Hospital Anxiety and Depression Scale (HADS)
Quality of sleep | Before and after the three months of interdisciplinary specialist interventions and after 12 months, which is standard procedure + after ending the add-on interventions and 24 months after the interdisciplinary treatments
  measured by Insomnia Severity Scale (ISI)

CONTACTS AND LOCATIONS:
Locations (1):
- Smärthjälpen, Gothenburg, Sweden